CLINICAL TRIAL: NCT04540679
Title: An Integrated Self-Management Service Delivery Model for Persons With SCI Across the Care Continuum
Brief Title: Self-Management Across the Care Continuum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: ForaHealthyMe Inc (Unknown); University Health Network, Toronto (Other); Spinal Cord Injury Ontario (Unknown); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Dalton Wolfe, Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 115501
Record Dates: First submitted 2020-08-25; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injuries
Keywords: online platform; self-management; e-health; care transitions
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: prospective experimental trial with two sets of participants a) Inpatients being randomized to one of two groups with pre-post assessments and b) outpatients being non-randomized with pre-post assessments
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inpatient - Standard Care Delayed Platform (Active Comparator): Patient will receive standard inpatient care and provided access to the platform 6 weeks after inpatient discharge with support provided by the VIP coach.
  Interventions: Other: VIP4SCI
- Inpatient - Platform Access (Active Comparator): Patient will be provided access to the platform within 2 weeks of admission to the inpatient program
  Interventions: Other: VIP4SCI
- Outpatient - Platform Access (Active Comparator): Patient will be provided access to the platform within 2 weeks of admission to the outpatient program. If patient is transitioning from the inpatient program, their access to the platform will be guided by which group they were originally assigned to (i.e. if a 6 week delay is applicable).
  Interventions: Other: VIP4SCI

INTERVENTIONS:
Other: VIP4SCI — Technology-enabled self-management & rehabilitation solution

SUMMARY:
Persons with spinal cord injury (SCI) face many challenges as they transition from inpatient care to outpatients and on into the community. With shorter lengths of stay and barriers to coordinating care between SCI specialists and community service providers, the development of self-management skills are an integral part in the effective community reintegration, proper healthcare utilization, management of secondary complications as well as independence and community participation. Based on the best available behaviour change theory, this initiative utilizes an online e-health Platform as a key component of a novel care service delivery model to enhance the development of effective self-management skills. This Platform will be provided to participants receiving care in the inpatient or outpatient programs at Parkwood Institute with the potential to continue its use in the community. Participants will complete surveys prior to, during and following use of the e-health solution. These will assess feasibility, usability, usage analytics and several patient-reported outcomes including self-management-related outcomes, healthcare utilization and prevalence of secondary complications. This platform is especially relevant to our current state of dealing with COVID-19 and the challenges it presents for clinicians and their patients in that it will provide an online solution during a time of physical isolation as well as providing access to tools and resources as people transition back to their home communities following specialized rehabilitation services.

DETAILED DESCRIPTION:
Participants using the e-health solution (called Parkwood VIP4SCI) will have access to features that connect them directly with their clinician(s) such as Virtual calling (initiated by the clinician), Messaging (email) and Scheduling/Calendar features. Platform use will be supported by a "VIP Coach. The clinician, coach and patient participants will also be able to use the e-health solution to create and monitor progress associated with self-management goals and also use embedded educational resources. These resources will also support the patients in best meeting their goals in a timely manner.

User Manuals for both the Client (i.e. Patient) and Provider (i.e. Clinician) are provided and contain screenshots and descriptive text that outline all the features of the intervention.

Patient participants will either be inpatients or outpatients, whereas healthcare team participants will consist of any provider assigned to the patient participant's circle of care at Parkwood Institute. The patient participants can choose to have their caregiver also access the platform - however, due to technical limitations, only 1 account is provided for the patient/caregiver dyad. Health care provider participants will have access to the platform for a specific patient at any time that patient is in the "Platform access" group as described below. The inpatient participants will be randomly allocated to 1 of 2 groups - either 1) "Platform access" or 2) "Standard care" with delayed access to the platform. In the "Standard care" group, the platform will be provided 6 weeks after inpatient discharge with support provided by the VIP coach. Those in the "Platform access" group will receive access within 2 weeks of admission to the inpatient or outpatient team at Parkwood Institute. For those patients transitioning from inpatient to outpatient care, their access to the platform will be guided by which group they were originally assigned to in addition to their needs and discharge circumstances as some of these patients may or may not be picked up by the Parkwood Outpatient team. The criteria influencing this will continue to be guided by the clinical team as per standard care. Participants seen by the outpatient team that were previously enrolled as inpatients in the "Standard care" group will be able to access the platform after 6 weeks of outpatient therapy with VIP coach support only, while those in the "Platform access" group can continue to use the platform with their outpatient health care providers.

Patient participants will complete surveys at specific time points throughout the study including measures at baseline (within 2 weeks of admission), discharge from inpatient program (or 6 weeks from admission for outpatients) and then 6 weeks after that. In the case of the "Standard care" group, there will be an additional follow-up survey to assess outcome measures 6 weeks after they have been provided access to the platform. The outcome measures will assess feasibility, usability, usage analytics and several patient-reported outcomes including self-management-related outcomes, healthcare utilization and prevalence of secondary complications.

ELIGIBILITY:
Inclusion Criteria - For patient participants:

* >18 years old
* Has a spinal cord injury
* Admitted to SCI inpatients/outpatients at Parkwood Institute for comprehensive Rehabilitation Care (not short stay)
* Has reliable high-speed internet access and device
* Intact cognitive function

Inclusion Criteria - For caregiver participants:

- Have been identified by the patient participant as someone who they would like to participate in a caregiver role

Inclusion Criteria - For health care provider participants:

- Part of the health care team for a patient participant

Exclusion Criteria - For patient participants only:

* <18 years old
* No spinal cord injury
* No access to reliable internet access or device
* Impaired cognitive function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-04-29 (Estimated); Study Completion 2021-04-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the use of the platform across 4 sub-domains including a) acceptance, b) demand, c) practicality, and d) limited efficacy | 6 weeks after admission/enrollment (inpatient/outpatient platform access groups), discharge (or 6 weeks after admission if outpatient), and 6 weeks after being provided access to the platform (if Standard Care group)
  Feasibility will be assessed across 4 subdomains (a) acceptance, b) demand, c) practicality, and d) limited efficacy) by the average scores from a set of 5 point likert-style questions relating to each sub-domain as part of a customized feasibility survey based on the Bowen et al feasibility framework (Am J Prev Med. 2009 May; 36(5): 452-457). The overall feasibility will be represented by the average score across all of the sub-domains.

SECONDARY OUTCOMES:
Social Roles & Activities - Ability to Participate | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using 4 questions from the Social Roles & Activities - Ability to Participate Short Form 10a which is a subscale in the SCI Quality of Life (SCI-QOL) 1.0 Measurement Tool (Tulsky et al., J Spinal Cord Med. May, 2015; 38(3): 257-269). This is a patient-reported outcome measure involving 5-point, likert-based questions.
Independence | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using 1 question from the Independence Short Form 8a which is a subscale in the SCI Quality of Life (SCI-QOL) 1.0 Measurement Tool (Tulsky et al., J Spinal Cord Med. May, 2015; 38(3): 257-269). This is a patient-reported outcome measure involving 5-point, likert-based questions.
Pressure Ulcer | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using 3 questions from the Pressure Ulcers Form 12a which is a subscale in the SCI Quality of Life (SCI-QOL) 1.0 Measurement Tool (Tulsky et al., J Spinal Cord Med. May, 2015; 38(3): 257-269). This is a patient-reported outcome measure involving 5-point, likert-based questions.
Pain Interference | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using 3 questions from the Pain Interference Form 10a which is a subscale in the SCI Quality of Life (SCI-QOL) 1.0 Measurement Tool (Tulsky et al., J Spinal Cord Med. May, 2015; 38(3): 257-269). This is a patient-reported outcome measure involving 5-point, likert-based questions.
Pain Behaviour | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using 1 question from the Pain Behaviour Form which is a subscale in the SCI Quality of Life (SCI-QOL) 1.0 Measurement Tool (Tulsky et al., J Spinal Cord Med. May, 2015; 38(3): 257-269). This is a patient-reported outcome measure involving 5-point, likert-based questions.
Resilience | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using 3 questions from the Resilience Short Form 8a which is a subscale in the SCI Quality of Life (SCI-QOL) 1.0 Measurement Tool (Tulsky et al., J Spinal Cord Med. May, 2015; 38(3): 257-269). This is a patient-reported outcome measure involving 5-point, likert-based questions.
Impact of Secondary Conditions | Longitudinal measure assessed at baseline and then at discharge (or 6 weeks) and then again 6 weeks later for follow-up
  This will be assessed using the Secondary Conditions Scale which involves 4-point, likert-based questions to indicate the degree to which a specific condition is a "problem" (Kalpakjian et al., J Spinal Cord Med. 2007; 30: 62-70). There are 16 questions, each one addressing a different condition (e.g., bowel dysfunction, bladder dysfunction, diabetes, etc) that are common in persons with spinal cord injury.
Quality of Mobile Application | 6 weeks after admission/enrollment (inpatient/outpatient platform access groups), discharge (or 6 weeks after admission if outpatient), and 6 weeks after being provided access to the platform (if Standard Care group)
  This will be assessed using the Mobile Application Rating Scale which is a series of 5-point likert-based questions across 6 sub-domains including (a) engagement, (b) functionality, (c) aesthetics, (d) information quality, (e) subjective quality and (f) perceived impact (Stoyanov et al., JMIR Mhealth Uhealth 2015;3(1):e27).

CONTACTS AND LOCATIONS:
Overall Officials: Dalton Wolfe, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No